CLINICAL TRIAL: NCT01113502
Title: A Phase I/II Study of Eltrombopag in Elderly Patients With AML
Brief Title: Eltrombopag in Elderly Acute Myelogenous Leukemia (AML)
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UPCC 17409
Record Dates: First submitted 2010-04-28; First posted 2010-04-30 (Estimated); Results first posted 2021-08-05 (Actual); Last update posted 2021-08-05 (Actual); Status verified 2021-07

CONDITIONS: Acute Myelogenous Leukemia (AML)
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — eltrombopag

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Phase 1 DL1 (Experimental): 50 mg; Taken daily by mouth
  Interventions: Drug: Eltrombopag
- Phase 1 DL 2 (Experimental): 100 mg; Taken daily by mouth
  Interventions: Drug: Eltrombopag
- Phase 1 DL3 (Experimental): 200 mg; Taken daily by mouth
  Interventions: Drug: Eltrombopag
- Phase 1 DL 4 (Experimental): 300 mg; Taken daily by mouth
  Interventions: Drug: Eltrombopag
- Phase 2 (Experimental): 200 mg taken daily by mouth for 2 weeks; then 300 mg taken daily by mouth
  Interventions: Drug: Eltrombopag

INTERVENTIONS:
Drug: Eltrombopag — Oral formulation taken daily
  Other Names: SB-497115-GR

SUMMARY:
This is a phase I/II open label study being conducted to evaluate the overall safety and initial effectiveness of an investigational drug, Eltrombopag in patients who are 60 years of age and older and who have Acute Myelogenous Leukemia (AML). Eltrombopag is an investigational drug, which means it has not been approved by the U.S. Food and Drug Administration (FDA) for use in this type of disease. Approximately 35 people will be enrolled on this study at the University of Pennsylvania

DETAILED DESCRIPTION:
Primary Objectives (Phase I Portion): 1). To determine the safety and tolerability of eltrombopag in elderly subjects with AML 2). To determine the maximally tolerated initial starting dose of eltrombopag for elderly subjects with AML Primary Objectives (Phase II portion): 1). To better define the safety and tolerability of eltrombopag in elderly patients with AML at the maximally tolerated starting dose Page 9 of 18 determined in Phase I portion of study. 2). To determine the incidence of peripheral platelet count improvement (using baseline and response parameters as defined below) for subjects with disease related thrombocytopenia. Secondary Objectives (Phase I and II): 1). To preliminarily determine the efficacy (using AML response criteria as defined below) of eltrombopag in elderly subjects with AML.

2). To perform ex-vivo analyses using subject AML samples and stock eltrombopag to 1) assess leukemic proliferative capacity and 2) investigate potential eltrombopag induced cytoxic mechanisms for leukemic cell death. 3). To perform pharmacodynamic assessments of drug activity in leukemic cells using subject samples collected at various time points before and during drug exposure. 4). To preliminarily correlate pharmacodynamic findings with clinical response.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of non-M3 AML which is either: a). Relapsed after standard chemotherapy or transplant;
* Newly diagnosed in a patient who is not an appropriate or willing candidate for standard induction chemotherapy - Age equal to or greater than 60 - Platelet count less than 75 - ECOG performance status of 0-2
* Life expectancy of at least 4 weeks
* Must be able to consume oral medication
* Must have recovered from toxic effects of prior chemotherapy
* Patients must be able to sign consent and be willing and able to comply with scheduled visits, treatment plan and laboratory testing.
* For Phase I portion only: Subject must be of non-East Asian (Japanese, Chinese, Taiwanese or Korean) descent.
* For Phase II portion subject can be either East Asian or non-East Asian descent.

Exclusion Criteria:

* Cytotoxic chemotherapy (including azacitidine or decitabine) within the past 28 days other than hydroxyurea
* Active participation in any other investigational treatment study for AML.
* Known HIV or Hepatitis C
* ECOG performance status greater than 2
* Uncontrolled intercurrent illness including, but not limited to: uncontrolled ongoing infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Previous therapy with romiplostim or any other TPO-R agonist

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2010-06 (Actual); Primary Completion 2013-03-14 (Actual); Study Completion 2015-11-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Noelle Frey, MD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I Dose Level I: 50 mg Eltrombopag taken daily by mouth
- Phase I Dose Level II: 100 mg Eltrombopag taken daily by mouth
- Phase I Dose Level III: 200 mg Eltrombopag taken daily by mouth
- Phase I Dose Level IV: 300 mg Eltrombopag taken daily by mouth
- Phase II Dose Level: 2 weeks of 200 mg Eltrombopag taken daily by mouth, then 300 mg Eltrombopag taken daily by mouth
Period: Overall Study
Arm/Group | Phase I Dose Level I | Phase I Dose Level II | Phase I Dose Level III | Phase I Dose Level IV | Phase II Dose Level
Started | 4 | 3 | 7 | 9 | 21
Completed | 3 | 3 | 3 | 6 | 21
Not Completed | 1 | 0 | 4 | 3 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 1 | 1 | 0
Not completed — Adverse Event | 0 | 0 | 3 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Phase I Dose Level I: 50mg Eltrombopag taken daily by mouth
- Phase I Dose Level II: 100mg Eltrombopag taken daily by mouth
- Phase I Dose Level III: 200mg Eltrombopag taken daily by mouth
- Phase I Dose Level IV: 300mg Eltrombopag taken daily by mouth
- Phase II: 2 weeks of 200mg Eltrombopag taken daily by mouth then 300mg Eltrombopag taken daily by mouth
- Total: Total of all reporting groups
Arm/Group | Phase I Dose Level I | Phase I Dose Level II | Phase I Dose Level III | Phase I Dose Level IV | Phase II | Total
Number analyzed (Participants) | 4 | 3 | 7 | 9 | 21 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 1 | 2 | 1 | 4 | 8
  >=65 years | 4 | 2 | 5 | 8 | 17 | 36
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2 | 4 | 8 | 16
  Male | 3 | 2 | 5 | 5 | 13 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 3 | 5 | 3 | 5 | 19
  Unknown or Not Reported | 1 | 0 | 2 | 6 | 16 | 25
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 2 | 1 | 1 | 4
  White | 4 | 3 | 4 | 7 | 11 | 29
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 1 | 1 | 9 | 11
Region of Enrollment [Number; unit: participants]
  United States | 4 | 3 | 7 | 9 | 21 | 44

OUTCOME MEASURES:

1. Primary Outcome: Maximally Tolerated Dose of Eltrombopag for Elderly Subjects With AML in Phase 1 Group
Description: The maximal tolerated dose of eltrombopag for elderly subjects with AML will be defined as the number of dose limiting toxicities per dosing level.
Time Frame: The time from first day of therapy until subject is off study treatment, an average of 10 weeks.
Measure: Number; unit: Dose Limiting Toxicities
Arm/Group | Phase I Dose Level I | Phase I Dose Level II | Phase I Dose Level III | Phase I Dose Level IV
Number analyzed (Participants) | 4 | 3 | 7 | 9
Dose Limiting Toxicities | 0 | 0 | 0 | 1
Statistical Analysis 1: Comparison: Phase I Dose Level I vs Phase I Dose Level II vs Phase I Dose Level III vs Phase I Dose Level IV; Test type: Other; Maximum Tolerated Dose (mg) = 300

2. Primary Outcome: Tolerability of Maximum Dose in Phase II Cohort
Description: The tolerability of eltrombopag in elderly patients with AML at the maximally tolerated starting dose determined in Phase I portion of study will be assessed by the number of dose limiting toxicities in the Phase II dosing cohort. Clinical assessment and laboratory evaluation of Adverse Events and DLTs will be done according to the Common Terminology Criteria for Adverse Events (CTCAE), version 4.0 of the National Cancer Institute (NCI) Cancer Therapy Evaluation Program (CTEP).
Time Frame: The time from first day of therapy to the first four weeks of therapy.
Measure: Number; unit: Dose Limiting toxicities
Arm/Group | Phase II Dose Level
Number analyzed (Participants) | 21
Dose Limiting toxicities | 0

3. Primary Outcome: The Safety of Eltrombopag for Elderly Subjects With AML in Phase 1 Group
Description: Safety of eltrombopag will be measured as the number of Grade 3 or higher adverse events per dosing level in Phase 1 group related to Eltrombopag. Relatedness is defined as event being assessed as unlikely, possibly, probably and definitely related to Eltrombopag. All events meeting these assessment categories will be considered related, and those assessed as Grade 3 or higher are reported for each dose level.
Time Frame: First day of study treatment to 30 days after last study treatment, an average of 10 weeks.
Measure: Number; unit: Related Adverse Events
Arm/Group | Phase I Dose Level I | Phase I Dose Level II | Phase I Dose Level III | Phase I Dose Level IV
Number analyzed (Participants) | 4 | 3 | 7 | 9
Related Adverse Events | 1 | 0 | 1 | 6

4. Primary Outcome: Safety of Eltrombopag in Patients With AML in Phase II Cohort.
Description: Safety of eltrombopag will be measured as the number of Serious Adverse Events in Phase II group related to Eltrombopag. Relatedness is defined as event being assessed as unlikely, possibly, probably and definitely related to Eltrombopag. All Serious Adverse Events meeting these assessment categories will be considered related and are reported for the Phase II cohort.
Time Frame: First day of study treatment to 30 days after last study treatment, an average of 7 weeks.
Measure: Number; unit: Number of related Serious Adverse Events
Arm/Group | Phase II Dose Level
Number analyzed (Participants) | 21
Number of related Serious Adverse Events | 0

5. Primary Outcome: Number of Participants With Peripheral Platelet Count Response in Phase I Cohort
Description: Peripheral platelet count response is defined by number of participants in each dosing cohort exhibiting a peripheral platelet count response using the IWG modified Hematologic Improvement response criteria: For patients with counts less than 100,000/ul: 1) For patients with baseline platelet of > 20,000/ul, absolute increase of platelet count by at least 30,000 /ul 2) For patients with baseline platelets < 20,000/ul, an increase to > 20,000/ul and by at least 100%.
Time Frame: First day of study treatment to 30 days after last study treatment, an average of 10 weeks.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I Dose Level I | Phase I Dose Level II | Phase I Dose Level III | Phase I Dose Level IV
Number analyzed (Participants) | 4 | 3 | 7 | 9
Participants | 0 | 0 | 2 | 2

6. Secondary Outcome: Overall Response Rate (Phase I and Phase II)
Description: This will include subjects who achieve a complete remission (CR) based on definitions by the International Working Group (IWG). CR is defined as the participant have a neutrophil Count>1000/ul, platelet count of >100,000/ul, bone Marrow Blasts < 5% and having no evidence of extramedullary disease.
Time Frame: The time from first day of therapy to time when subject achieves a complete remission (CR), based on the definition of the International Working Group (IWG), approximately 30 days.
Measure: Number; unit: Participants with a CR
Arm/Group | Phase I Dose Level I | Phase I Dose Level II | Phase I Dose Level III | Phase I Dose Level IV | Phase II Dose Level
Number analyzed (Participants) | 4 | 3 | 7 | 9 | 21
Participants with a CR | 0 | 0 | 0 | 1 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were collected on each subject from the time of treatment initiation until 30 days after the last treatment administration, an average of 14 weeks for the Phase I cohort, and an average of 11 weeks for the Phase II cohort.
Description: Adverse event data for the total counts of the Phase II cohort is available, but the number of individual events per participant in this dosing group is not available. These data have been searched for in all the available reports and materials, requested from the PI, requested from institutional leadership, searched for in institutional clinical trial databases and medical records, but cannot be located.
Arm/Group | Phase I Dose Level I | Phase I Dose Level II | Phase I Dose Level III | Phase I Dose Level IV | Phase II Dose Level
All-Cause Mortality (participants affected / at risk) | 2/4 | 1/3 | 3/7 | 2/9 | 0/21
Serious Adverse Events (participants affected / at risk) | 3/4 | 3/3 | 7/7 | 7/9 | 9/21
Other Adverse Events (participants affected / at risk) | 2/4 | 0/3 | 3/7 | 5/9 | 0/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I Dose Level I (N=4) | Phase I Dose Level II (N=3) | Phase I Dose Level III (N=7) | Phase I Dose Level IV (N=9) | Phase II Dose Level (N=21)
Blood and lymphatic system disorders - Other, Specify (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — hospitalization for clot in PICC line
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (3) | 1 (1) | 3 (4) | 2 (2) | 3 (4)
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) — Lung cancer
Death, NOS (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — Hospitalization due to progressive disease
Fatigue (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intracranial hemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Neck edema (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anorexia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Disease progression (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fever (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anorectal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombocytopenia (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bronchial Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I Dose Level I (N=4) | Phase I Dose Level II (N=3) | Phase I Dose Level III (N=7) | Phase I Dose Level IV (N=9) | Phase II Dose Level (N=21)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 3 | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain, abdominal (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
White blood cell decrease (Investigations) | 1 (1) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Aspiration Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Activated PTT prolongation (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)

LIMITATIONS AND CAVEATS:
Adverse event data for the total counts of the Phase II cohort is available, but the number of individual events per participant in this dosing group is not available. These data have been searched for in all the available reports and materials, requested from the PI, requested from institutional leadership, searched for in institutional clinical trial databases and medical records, but cannot be located.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes